CLINICAL TRIAL: NCT03877250
Title: Characterization of Mechanism of Response to PD-1 Blockade in NSCLC: A Pilot Study
Brief Title: Analysis of Biopsy Specimens to Study Responses to PD-1 or PD-L1 Therapies
Status: Withdrawn | Type: Observational
Why Stopped: The primary objectives have not been met due to no patient enrollment therefore, the PI is requesting to close the study at this time.
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Wang Initiative in Lung Cancer Clinical Trials (Unknown)
Responsible Party: Sponsor
Other Study IDs: 19-030
Record Dates: First submitted 2019-03-12; First posted 2019-03-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2020-08

CONDITIONS: Non Small Cell Lung Cancer
Keywords: PD-L1 High; 19-030; Memorial Sloan Kettering Cancer Center
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Device: No

GROUPS / COHORTS (1):
- Non Small Cell Lung Cancer (NSCLC): Participants with pathologically confirmed newly diagnosed or recurrent advanced NSCLC that is PD-L1 high by immunohistochemistry
  Interventions: Diagnostic Test: Pre-Treatment Biopsy; Diagnostic Test: On-Treatment Biopsy; Diagnostic Test: Biopsy at Disease Progression; Diagnostic Test: Peripheral Blood-Based Studies

INTERVENTIONS:
Diagnostic Test: Pre-Treatment Biopsy — Participants screened for participation will include those with a diagnosis of advanced NSCLC who have undergone a pre-treatment biopsy prior to start of therapy with a PD-(L)1 inhibitor or who are medically able to undergo a biopsy if (1) no pre-treatment biopsy has been obtained and (2) no PD-(L)1 inhibitor has been started.
Diagnostic Test: On-Treatment Biopsy — All participants who receive at least 1 dose of PD-(L)1 inhibitor will be referred for a biopsy. The biopsy should be obtained within 4 weeks of first on-treatment imaging (usually performed ~6-9 weeks after beginning therapy) and will be performed in participants regardless of radiologic response.
Diagnostic Test: Biopsy at Disease Progression — All participants who develop disease progression after initial response to PD-(L)1 blockade will be considered for an additional, optional biopsy. Biopsies at disease progression are often obtained per standard of care within 4 weeks of documented progression on imaging and prior to the initiation of further systemic therapy.
Diagnostic Test: Peripheral Blood-Based Studies — All participants will have peripheral blood obtained on Day 1 of cycles 1-4 (0, 3, 6, and 9 weeks). At each time point, peripheral blood sample will be collected pre-treatment and used for analysis of T cell subsets and TCR sequencing.

SUMMARY:
The purpose of this study is to attempt to obtain an on-treatment biopsy in participants with non-small cell lung cancer who are receiving standard treatment with a drug that targets the PD-1 or PD-L1 protein.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed newly diagnosed or recurrent advanced Non Small Cell Lung Cancer/NSCLC that is PI-L1 high by immunohistochemistry (PD-L1 >/= 50%)
* Intended treatment with a PD-(L)1 inhibitor
* Age >/= 18 years
* Karnofsky Performance Status >/= 70% and medically fit to undergo a biopsy procedure

Exclusion Criteria:

* Any medical condition or any sites of disease that would preclude a biopsy
* Pregnant or breastfeeding women
* Cognitively impairment affecting ability to understand and provide informed consent
* Prior PD-(L)1 blockade treatment
* Chemotherapy within 6 months prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with newly diagnosed or recurrent, PD-L1 high (>50%) metastatic non-small cell lung cancer without prior PD-(L)1 therapy
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-03-08 (Actual); Primary Completion 2020-08-26 (Actual); Study Completion 2020-08-26 (Actual)

PRIMARY OUTCOMES:
Number of participants biopsied on-treatment and with newly diagnosed or recurrent PD-L1 advanced Non Small Cell Lung Cancer/NSCLC | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Hellmann, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (6):
- United States (6):
  - Memoral Sloan Kettering Basking Ridge (Consent and Follow up), Basking Ridge, New Jersey
  - Memoral Sloan Kettering Monmouth (Consent and Follow up), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Consent and Follow up), Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk (Consent Only), Commack, New York
  - Memoral Sloan Kettering Westchester (Consent & Follow Up), Harrison, New York
  - Memorial Sloan - Kettering Cancer Center (Consent and follow-up), New York, New York

IPD SHARING:
Plan to Share IPD: Yes
• Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org